CLINICAL TRIAL: NCT04996251
Title: Clinical Effectiveness of Pre-incision Versus Post-incision Local Anesthetic During Laparoscopic/Robotic Sacrocolpopexy
Brief Title: Pre-incision Versus Post-incision Local Anesthetic During Robotic Sacrocolpopexy
Acronym: CLAPPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Harvey Winkler, MD, System Chief of Urogynecology Division; Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-0422
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- subcutaneous infiltration pre-incision (Experimental): Marcaine (bupivacaine) injected in the umbilical port site subcutaneously, while in the other 4 sites injection under direct visualization
  Interventions: Drug: Bupivacaine Injection
- subcutaneous infiltration post-incision (Experimental): local anesthetic infiltrated subcutaneously at the end of the procedure after trocar removal and after skin closure with suture
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — 0.25% Bupivacaine being used as local anesthetic to inject into incision sites of tracer sites during a laparoscopic/robotic-assisted sacrocolpopexy
  Other Names: Marcaine

SUMMARY:
Obtaining Likest-pain scale score on postoperative day one after injection of local anesthetic into incision sites of a laparoscopic/robotic-assisted sacrocolpopexy

DETAILED DESCRIPTION:
Pelvic organ prolapse is becoming more common as women's life expectancy is increasing and the prevalence of obesity is rising. Many women undergo pelvic reconstructive surgery to treat their prolapse and improve their quality of life. The incidence of pelvic organ prolapse is 1.5-1.8 surgeries per 1,000 women years. Approximately 300,000 pelvic reconstructive surgeries are performed each year in the United States. There is a wide variety in surgical approaches and procedures for prolapse. One such procedure is a sacrocolpopexy in which the cervix or vaginal cuff is lifted to the anterior longitudinal ligament overlying the sacrum via a mesh graft. This can be done in a minimally invasive fashion with a laparoscopic or robotic approach or in an open abdominal approach. Numerous studies have shown this procedure to have a high success rate and long-term durability. As robotic/laparoscopic approach to surgery has shown shorter hospital-stays and improved patient outcomes, the robotic-assisted sacrocolpopexy has been rapidly incorporated into clinical practice.

In general, surgery causes a release of painful chemical mediators which has led to increased narcotic use, increased narcotic addiction, and number of pills prescribed. Most individuals who undergo surgery will require narcotics postoperatively to control their pain and some individuals have to extend their hospital stay until adequate pain control is achieved. Our study is aimed to reduce narcotic use, decrease hospital stay due to pain issues and determine if timing of adjunct pain medication improves pain scales for patients.

As postoperative pain after minimally invasive surgery is complex, specialists suggest that the effective analgesic treatment should be a multimodal approach. Use of local anesthetic with bupivacaine at robotic/laparoscopic trocar sites is the standard of care, however, there is no standard as to optimal timing that is most beneficial for patients to decrease pain. Currently, bupivacaine is used by providers at the trocar sites at either the beginning of the case or at the end of the case. From clinical observation, it appears that postoperative pain levels reported from patients receiving either at the beginning of surgery (pre-) or end (post-incision) of the surgery are similar. This study aims to examine the difference in postoperative day one pain levels reported by patients between the two infiltration methods

ELIGIBILITY:
Inclusion Criteria:

* Females 18+ years old who are undergoing robotic/laparoscopic assisted sacrocolpopexy

  * With/without hysterectomy
  * With/without unilateral/bilateral salpingectomy
  * With/without unilateral/bilateral oophorectomy
  * With/without mid-urethral sling
  * With/without anterior/posterior vaginal repair

    * English or Spanish speaking
    * Weight ≥ 120 lb

Exclusion Criteria:

* Females < 18 years old

  * Chronic pelvic pain/chronic pain syndromes
  * Fibromyalgia
  * Pregnant or breastfeeding patients
  * Concomitant procedure for hernia repair or rectal prolapse repair
  * Undergoing primary vaginal prolapse surgery
  * Contraindications to taking the following medications: Bupivacaine
  * Patients who weight is < 120lb
  * Hypersensitivity to bupivacaine hydrochloride, amide-type local anesthetics, or any component of the formulation
  * Pudendal or spinal nerve block given during surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) with any other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Infiltration Pre-incision | Subcutaneous Infiltration Post-incision
Started | 62 | 67
Completed | 62 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Infiltration Pre-incision | Subcutaneous Infiltration Post-incision | Total
Number analyzed (Participants) | 62 | 67 | 129
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [57.8 to 66] | 62 [53.3 to 67.8] | 62 [53.3 to 67.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Total number of patients participating [Count of Participants; unit: Participants] | 62 | 67 | 129

OUTCOME MEASURES:

1. Primary Outcome: Likert-pain Scale Score on Postoperative Day One
Description: Difference in Likert-pain scale score difference between pre-incision versus post-incision subcutaneous infiltration with 4-5 milliliters 0.25% Bupivacaine (0 is no pain; 10 is worst pain imaginable)
Time Frame: 18-24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subcutaneous Infiltration Pre-incision | Subcutaneous Infiltration Post-incision
Number analyzed (Participants) | 62 | 67
units on a scale | 2.94 (2.36) | 3.27 (2.33)

2. Secondary Outcome: Narcotic Usage
Description: Compare narcotic usage (pills used) until first postoperative appointment
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Subcutaneous Infiltration Pre-incision | Subcutaneous Infiltration Post-incision
Number analyzed (Participants) | 62 | 67
MME | 0 [0 to 16.9] | 0 [0 to 22.5]

ADVERSE EVENTS:
Time Frame: 23 months
Arm/Group | Subcutaneous Infiltration Pre-incision | Subcutaneous Infiltration Post-incision
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/67
Other Adverse Events (participants affected / at risk) | 0/62 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT04996251/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT04996251/ICF_001.pdf